CLINICAL TRIAL: NCT05125523
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Antitumor Activity of Sirolimus for Injection (Albumin Bound) in Patients With Advanced Solid Tumors
Brief Title: A Study of Sirolimus for Injection (Albumin Bound) in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1901-CSP-001
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumors
Keywords: Sirolimus for Injection (Albumin Bound)
MeSH Terms: interventions — Sirolimus; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus for Injection (Albumin Bound) (Experimental): Stage 1：Multiple doses of Sirolimus for Injection (Albumin Bound) will be administered intravenously.
  Stage 2：RP2D of Sirolimus for Injection (Albumin Bound) as determined during stage 1 will be administered intravenously.
  Interventions: Drug: Sirolimus for Injection (Albumin Bound)

INTERVENTIONS:
Drug: Sirolimus for Injection (Albumin Bound) — Sirolimus for Injection (Albumin Bound), intravenously, once a week, 28 days per cycle (three weeks-on and one week-off)

SUMMARY:
The purpose of this study is to estimate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of Sirolimus for Injection (Albumin Bound) in patients with solid malignancies.

DETAILED DESCRIPTION:
This study will be conducted in two stages.

Stage 1: To evaluate the safety and tolerability of Sirolimus for Injection (Albumin Bound) in patients with advanced tumors, determine the MTD and RP2D. The dose escalation scheme using the accelerated titration design for dose 1 and the rolling-six design for the remaining doses.

Stage 2: To preliminarily assess the antitumor activity of Sirolimus for Injection (Albumin Bound). Patients will be assigned to different cohorts based on their tumor type.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (inclusive), no gender limitation.
2. Patients must have a histologically or cytologically confirmed advanced or metastatic tumor for which no effective standard therapy is available, or have failed or been intolerant to standard therapies.
3. At least one measurable lesion per RECIST version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
5. Life expectancy of ≥3 months.
6. Suitable organs and hematopoietic function should be available. Laboratory tests during screening should meet the appropriate criteria.
7. Signed informed consent form.

Exclusion Criteria:

1. Prior anticancer treatment or participation in another clinical study within 4 weeks (or 5 half-lives of the treated drug, whichever is longer) prior to the first dose of study drugs.
2. Patients who have undergone major surgery within 4 weeks prior to starting study treatment, or who have not fully recovered from previous surgery.
3. Unresolved toxicities from prior therapy greater than Grade 1 as per Common Terminology Criteria for Adverse Events (CTCAE) (except alopecia or any other toxicity without safety risks as judged by the investigator).
4. History of serious cardiovascular disease.
5. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, and the investigator judges it to be unsuitable for inclusion.
6. Known prior hypersensitivity to study drugs or any component in their formulations.
7. Prior treatment with any mTOR inhibitor.
8. Has received a live or live-attenuated virus vaccine within 30 days prior to consent.
9. Uncontrollable active infection (CTCAE v5.0 ≥grade 2).
10. Use of strong inhibitors and inducers of CYP3A4 within 2 weeks prior to receiving the first dose of study drug and still need to continue using this class of drug.
11. History of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency, or organ transplant history.
12. HBsAg-positive with HBV viral load (VL) ≥1000 IU/mL; Hepatitis C Virus (HCV)-positive; Anti-treponema pallidum positive.
13. Women of child-bearing potential, or men whose partners are women of childbearing age, have not agree to use highly effective methods of contraception during dosing and for 6 months after study drug discontinuation; female patients has a positive serum pregnancy test within 7 days prior to receiving the first dose of study medication; lactating female.
14. Has history of other serious diseases judged by the investigator, which will threaten the safety of patients or interfere the study compliance, or other reasons are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 3 years
Dose-Limiting Toxicities (Stage 1) | Cycle 1 (Up to 28 days)
Maximum tolerated dose (Stage 1) | Up to 1.5 years
Recommended phase 2 dose (Stage 1) | Up to 1.5 years
Overall response rate (Stage 2) | Up to 3 years

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Peak concentration (Cmax) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Peak time (Tmax) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Distribution volume (Vz) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Elimination half-life (t1/2) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Clearance (CL) | Day 1 of cycle 1 to Day 1 of cycle 4 (85 days)
Disease Control Rate | Up to 3 years
Duration of Response | Up to 3 years
Progression-free Survival | Up to 3 years
4ebp-1 phosphorylation level in blood samples | Up to 168 hours post dose
S6K phosphorylation level in blood samples | Up to 168 hours post dose
TSC1/2 status in tumor samples | Day 1 of cycle 1
PTEN status in tumor samples | Day 1 of cycle 1
PIK3CA status in tumor samples | Day 1 of cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No